CLINICAL TRIAL: NCT01431690
Title: An Open-label, 2-cohort Study to Evaluate the Effect of Multiple Doses of Epanova® on the Single Dose Pharmacokinetics and Pharmacodynamics of Warfarin and to Compare the Systemic Exposure of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) Following Multiple-dose Administrations of Epanova® Compared to Lovaza® in Healthy Normal Subjects
Brief Title: Interaction of Epanova on Warfarin Pharmacokinetic and Anticoagulant Activity and Comparison of the Effects of Epanova and Lovaza on Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) After Low-fat Meals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OM-EPA-006
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Hypertriglyceridemia
Keywords: Eicosapentaenoic Acid; Docosahexaenoic Acid; Warfarin; Hypertriglyceridemia; Omega-3 free fatty acids; Omega-3 ethyl ester acids; Epanova; Lovaza; pharmacokinetics; low-fat meal
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Warfarin; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin and Epanova (Experimental)
  Interventions: Drug: warfarin; Drug: omefas
- Lovaza (Active Comparator)
  Interventions: Drug: omega-3-acid ethyl esters

INTERVENTIONS:
Drug: warfarin — A single 25 mg dose of warfarin
  Other Names: coumarin-based anticoagulant
  Arms: Warfarin and Epanova
Drug: omefas — 4 x 1 g capsule dose of Epanova®
  Other Names: Epanova
  Arms: Warfarin and Epanova
Drug: omega-3-acid ethyl esters — 4 x 1 g capsule dose of Lovaza®
  Other Names: Lovaza
  Arms: Lovaza

SUMMARY:
The primary objective of this study is to determine the effect of Epanova® on the pharmacokinetic and anticoagulant activity of warfarin.

The secondary objective of this study is to compare the systemic exposure of EPA and DHA following multiple-dose administration of Epanova®, a free fatty acid mixture, to Lovaza®, a mixture of fatty acid ethyl esters, under low-fat meal conditions since these products are likely to be administered to patients with cardiovascular disease who are recommended to consume low-fat meals.

ELIGIBILITY:
Inclusion Criteria:

Subject candidates must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Healthy adult male and/or females, 18 to 55 years of age (inclusive).
2. Body mass index (BMI) ≥ 18 and ≤ 29.9 (kg/m2).
3. Medically healthy with clinically insignificant screening results. Hemoglobin must be ≥ the lower limit of normal.
4. Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to dosing.
5. Voluntarily consent to participate in the study and to follow the restrictions and procedures outlined for the study.
6. For the Warfarin and Epanova Arm, females must be of non-childbearing potential defined as have undergone sterilization procedures at least 6 months prior to check-in or have been postmenopausal for at least 24 consecutive months prior to check-in of the study and have a screening follicle stimulating hormone level > 40 mIU/mL.
7. For the Lovaza Arm, females may be of non-childbearing potential (as outlined above for Warfarin and Lovaza) or be of childbearing potential and must either be sexually inactive (abstinent) for 14 days prior to screening and remain so through 30 days following the final dosing of the study drug or until completion of the subject's first menstrual cycle following the final dosing of the study drug, whichever period of time is longer or have been using one of the acceptable methods of birth control.

Exclusion Criteria:

Subjects may be excluded from the study if there is evidence of any of the following criteria at screening, check-in, or at any time during the study as appropriate.

For both arms (Warfarin and Epanova, Lovaza)

1. Has a history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Has a positive urine drug/alcohol testing at screening or check-in.
3. Has a positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
4. Has consumed fish within 7 days prior to check-in.
5. Has used fish oil, other EPA and/or DHA containing supplements within 2 months of check-in.
6. Has a history or presence of alcoholism or drug abuse within the 2 years prior to check-in.
7. Has a known sensitivity or allergy to soybeans, fish, and/or shellfish.
8. Has had a hypersensitivity or idiosyncratic reaction to compounds related to Epanova® and Lovaza®.
9. Has used any prescription medication (with the exception of hormonal contraceptives for females in the Lovaza arm) within 14 days prior to check-in.
10. Has used any over-the-counter (OTC) medication, including herbal products (e.g., bromelains, danshen, dong quai [Angelica sinesis], garlic, ginko biloba, ginseng, and St. John's wort), within the 7 days prior to check-in. Up to 2 g per day of acetaminophen is allowed at the discretion of the PI for the Lovaza arm.
11. Has used any drugs known to significantly inhibit [strong or moderate] or induce liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to check-in.
12. Has donated blood or has had a significant blood loss within 56 days prior to check-in.
13. Has donated plasma within 7 days prior to check-in.
14. Has participated in another clinical trial within 30 days prior to check-in.
15. Is a female who is pregnant or lactating.

For Warfarin and Epanova Arm only:

1. Has taken large daily doses of Vitamin K (exceeding 25 μg/day) or has eaten large quantities (e.g., averaging > 4 portions daily) of dark green/leafy vegetables (e.g., spinach, kale, collard greens, broccoli, Brussels sprouts) during the 2 months prior to check-in.
2. Is employed or involved in any circumstance which would place them at increased risk of hemorrhage (e.g., contact sports, strenuous or unaccustomed weight lifting, running, bicycling).
3. Has a personal or familial history of bleeding disorder(s), thromboembolic disease, clinical GI bleeding, or any history of GI surgery except uncomplicated appendectomy or cholecystectomy, or colorectal surgery for polyps, nonmalignant tumors, or diverticula.
4. Has active severe gingivitis.
5. Has had a hypersensitivity or idiosyncratic reaction to compounds related to warfarin.
6. Has a recent physical injury (within the 2 weeks prior to screening).
7. Has had a major surgery within the 3 months prior to screening.
8. Is allergic to Vitamin K.
9. Has used non-steroidal anti-inflammatory (NSAID) drugs within the 2 weeks prior to check-in.
10. Has a positive fecal occult blood sample at check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of R- and S- warfarin | 168 hours
  The primary endpoints of this study will be the area under the curve (AUC)0-t, AUC0-inf, and maximum concentration (Cmax) of R- and S warfarin and the maximum International Normalized Ratio (INRmax) over 168 hours postdose and INR AUC0-168 when warfarin is administered with and without Epanova®.
Pharmacodynamics of R- and S- warfarin | 168 hours
  The INRmax over 168 hours postdose and INR AUC0-168 when warfarin is administered with and without Epanova®.

SECONDARY OUTCOMES:
Total EPA+DHA | 24 hours
  The AUC0-tau and Cmax of baseline-adjusted total EPA+DHA following multiple doses (14 days) of Epanova® and Lovaza®.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, FACC, Study Director — Omthera Pharmaceuticals, Inc
Locations (1):
- Tempe, Arizona, United States